CLINICAL TRIAL: NCT04457791
Title: Improving Constipation by Stimulating Fiber Intake Using Personalized Dietary Advice
Acronym: PAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Maag Lever Darm Stichting (Other); TNO (Other); Sensus (Industry); Kellogg Company (Industry); Bolletje (Unknown); Sonneveld (Unknown); Roquette Freres (Industry); Nederlands Bakkerij Centrum (Other); Wageningen Food and Biobased Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NL73256.028.20
Record Dates: First submitted 2020-06-18; First posted 2020-07-07 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Constipation
Keywords: Dietary fiber; Personalized advice
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: One group is followed over time (within person design)
Who Masked: Participant
Masking Description: participants are not informed about the content and focus of the personalized dietary advice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention phase (Experimental): From week 5-8, participants will receive the intervention, namely personalized dietary advice.
  Interventions: Behavioral: Personalized dietary advice
- Observational phase (No Intervention): From week 1-4, participants will not receive any intervention, but just will be observed, to form as their own control

INTERVENTIONS:
Behavioral: Personalized dietary advice — Via an self-developed website and algorithm, participants will receive digital personalized dietary advice to increase dietary fiber intake, aiming to reduce constipation complaints. The advice is personalized on phenotype (habitual diet, gender)
  Arms: Intervention phase

SUMMARY:
Rationale: constipation-related complaints are prevalent in 5-20% of the population.

Dietary fibers play a crucial role in improving and maintaining gut health, increasing stool weight, stool frequency and improvement of stool consistency. Currently, very few adults meet the recommendation of 30 (females) or 40 (males) grams of fiber per day. Personalized dietary advice may be the solution to increase dietary fiber intake and reduce constipation-related complaints in large populations. Objective: To investigate the effectiveness of personalized dietary advice (PDA) in reducing constipation-related complaints, by increasing dietary fiber intake in people with constipation-related complaints. Study design: This study has a one-group pre-test post-test design with a run-in period.

The duration of the study is 8 weeks, which includes a 4-week run-in phase and a 4-week intervention period. All subjects receive the PDA. Study population: adult subjects with constipation-related complaints, defined as predominant Bristol stool form between 1-4 and not satisfied with their bowel habits (scale ranging from 1-10, cut-off <6). Possibly stool frequency ≤4 stools per week will be included as a definition. Subjects need to have a relatively low dietary fiber intake defined as <26 grams (females) or <33 grams (males), which is ≥15% below the recommendation of fiber intake. Intervention: personalized advice based on their habitual food pattern (as assessed using a food frequency questionnaire) and preferences. Based on a special algorithm, the PDA provides high fiber alternatives for low-fiber products that subjects currently use, close to their current eating behavior, to help increase dietary fiber intake. This PDA will be provided using an online web-portal.

Main study parameters/endpoints:primary outcomes are stool pattern, gastrointestinal complaints and constipation quality of life and severity. Secondary parameters include dietary fiber intake, physical activity, body weight, psychological questionnaires, and fecal microbiota composition and metabolite levels. Furthermore, the PDA will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 55 years
* BMI <30 kg/m2
* Has constipation related complaints: response <6 to the question "how satisfied are you with your stool pattern", which is rated on a visual analog scale (VAS) from 1-10, together with at least one of the following criteria:

  1. Habitual stool form of Bristol stool type 1-4 or
  2. ≤4 defecations per week
* living in the surroundings of wageningen (max. 50km)
* in possession of a computer with chrome browser and a mobile phone compatible with applications Note: these criteria are less stringent than the official "constipation" definition, because we preferably want to include participants that do not use laxatives (yet), and we assume that in this 'mild constipation' group increasing fiber intake can have the most beneficial effects. Moreover, we chose not to use the Rome IV criteria as definition of constipation-related complaints, due to the proven inability to distinguish functional constipation from Irritable Bowel Syndrome. If there are sufficient eligible participants, the participants with the lowest stool frequency will be selected
* Relatively low fiber intake (females <26 grams, males <33 grams). When enough eligible participants are available, we will choose the participants with the lowest dietary fiber intake.
* signed informed consent

Exclusion Criteria:

* Subjects with a disease that may interfere with the personal dietary advice or outcomes, such as a known autonomic disorder, inflammatory bowel disease, coeliac disease, cancer, dialysis patients, chronic kidney failure, depression or hypothyroidism.
* Currently following strict diet and unwilling or unable to change; for example a gluten free diet or a "crash diet" using meal substitutes
* Use of medication that can interfere with the study outcomes, including diuretics, antidepressants, codeine, antibiotics or fiber supplements. Preferably laxative use is excluded, but if recruitment is hurdled by this, we at least exclude specific laxatives like resolor, relistor and constella. These are laxatives who have a significant impact on bowel movements, and are only available on prescription. Osmotic (over the counter available) laxatives will be included if recruitment is difficult. Subjects will then be asked to keep their laxative use stable or reduce, but not to increase usage from their habitual pattern (unless necessary, but then report it to the researchers). Moreover, additional questions regarding laxative usage will be included to estimate the effect of laxatives on stool pattern.
* Female subjects: currently pregnant or breastfeeding, or intending to become pregnant during the study, as this can affect stool patterns and wellbeing.
* Are simultaneously participating in another study.
* Unwilling or unable to fulfil the study criteria.
* Student or employee working at Food, Health and Consumer Research from Food and Biobased Research, or Department of Human Nutrition & Health, Wageningen University.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Change in constipation severity after 8 weeks | Measured during week 1, week 4 and week 8
  Will be measured using a validated questionnaire PAC-SYM, which has 12 items. Scores can range between 1 (not severe) and 4 points (vere severe)
Change in constipation related quality of life after 8 weeks | Measured during week 1, week 4 and week 8
  Will be measured using a validated questionnaire (PAC-QoL), which has 28-items
Stool pattern | 8 weeks
  Will be assessed daily using a mobile phone application (using ecogological momentary assessment, EMA). Subjects will indicate each day whether they had defecation and which type of defecation it was (based on the bristol stool chart)
Abdominal pain | 8 weeks
  Measured daily using a mobile phone application EMA, on a 10-point visual analog scale rangeing from not at all to very severe
Bloating | 8 weeks
  Measured daily using a mobile phone application EMA, on a 10-point visual analog scale rangeing from not at all to very severe
Flatulence | 8 weeks
  Measured daily using a mobile phone application EMA, on a 10-point visual analog scale rangeing from not at all to very severe
Fatigue | 8 weeks
  Measured daily using a mobile phone application EMA, on a 100-point visual analog scale rangeing from not at all to very severe
Abdominal cramps | 8 weeks
  Measured daily using a mobile phone application EMA, on a 10-point visual analog scale rangeing from not at all to very severe

SECONDARY OUTCOMES:
Dietary fiber intake | during week 1, week 4 and week 8 of the study
  Measured by 24hr recall. Each measurement will consist of 3 days to take variance into account (1 weekend day and 2 weekdays)
Short fiber screening questionnaire | At screening
  Validation of a short fiber screening questionnaire: 18-item questionnaire assessing fiber intake
Laxative use | Daily during 8 weeks
  Measured daily using a mobile phone application EMA: did you use laxatives today. If yes: which laxative
Physical activity level | during week 1, week 4 and week 8
  Will be measured by the validated short questionnaire to assess health-enhancing physical activity (SQUASH)
Body weight | During week 1, week 4 and week 8
  Measured during study visits on a weighing scale
Microbiota composition from fecal samples, as assessed by 16S rRNA sequencing | During week 1, week 4, and week 8
  Will be measured from fecal samples taken by participants' at home
short-chain fatty acid levels from fecal samples, assessed by HPLC | During week 1, week 4 and week 8
  Will be measured from fecal samples taken by participants' at home
Validated subjective health questionnaire | During week 1, week 4 and week 8
Self-regulation questionnaire | During week 1, week 4 and week 8
intention to eat fibers questionnaire | During week 1, week 4 and week 8
subjective knowledge of fibers questionnaire | During week 1, week 4 and week 8
outcome beliefs of fibers questionnaire | During week 1, week 4 and week 8
self-efficacy of fiber intake | Daily during the intervention period of 4 weeks
  Measured by the question: did you manage to eat more fiber today: on a 100-point visual analog scale from "not at all" to "yes, completely" using a mobile phone application on the phone
Evaluation questionnaire | During week 8
  That evaluates the personalized dietary advice

CONTACTS AND LOCATIONS:
Overall Officials: Nicole de Wit, PhD, Principal Investigator — Wageningen Food and Biobased Research
Locations (1):
- Wageningen University & Research, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rijnaarts I, de Roos N, Zoetendal EG, de Wit N, Witteman BJM. Development and validation of the FiberScreen: A short questionnaire to screen fibre intake in adults. J Hum Nutr Diet. 2021 Dec;34(6):969-980. doi: 10.1111/jhn.12941. Epub 2021 Aug 29. PMID 34378249